CLINICAL TRIAL: NCT00137345
Title: A Randomized, Open-Label, Comparative Evaluation of the Safety and Efficacy of Sirolimus Versus Cyclosporine When Combined in a Regimen Containing Basiliximab, Mycophenolate Mofetil, and Corticosteroids in Primary De Novo Renal Allograft Recipients
Brief Title: Study Comparing Sirolimus With Cyclosporine in a Calcineurin Inhibitor (CNI)-Free Regimen in Kidney Transplant Recipients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468H1-318; B1741188 (Other: Pfizer)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2006-09

CONDITIONS: Kidney Transplant
Keywords: Randomized controlled trial; Clinical Trial Phase III; Drug therapy; Immunosuppression; Treatment outcome; Kidney transplantation; Kidney function tests
MeSH Terms: interventions — Sirolimus

INTERVENTIONS:
Drug: sirolimus

SUMMARY:
The purpose of this study is to determine if one drug is superior to another with regard to safety and the preservation of renal function after a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis patients who will be receiving their first kidney transplant
* Weight over 88 pounds (lbs.)

Exclusion Criteria:

* Very high cholesterol levels
* Obesity
* Organ donor over 65 years of age if living; over 60 years of age if cadaveric.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 2005-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To demonstrate the superiority of the sirolimus regimen versus cyclosporin A by intent to treat analysis of kidney function at 52 weeks, measured by mean glomerular filtration rate (GFR)
Non-inferiority of the composite of graft loss and death at 52 weeks

SECONDARY OUTCOMES:
Incidence and severity of rejection at 12, 24, 52, 104, 156, 208 weeks; GFR at 24, 104, 156, 208 weeks; progression of chronic allograft nephropathy or deterioration of transplanted kidney at 52 weeks
quality of life at 24, 52 and 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, MedInfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Norway, Sweden, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For Australia, Taiwan, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Austria, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Italy, Greece, decresg@wyeth.com; Trial manager, Principal Investigator — For Hungary, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For Turkey, Erisc@wyeth.com; Trial Manager, Principal Investigator — For South Africa, ZAFinfo@wyeth.com; Trial Manager, Principal Investigator — For Argentina, Chile, scheima@wyeth.com, rendop@wyeth.com; Trial Manager, Principal Investigator — For UK, ukmedonfo@wyeth.com; Trial Manager, Principal Investigator — For Switzerland, med@wyeth.com
Locations (73):
- United States (21):
  - San Diego, California
  - San Francisco, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Gainesville, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Portland, Maine
  - Springfield, Massachusetts
  - Detroit, Michigan
  - New York, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Toledo, Ohio
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Dallas, Texas
  - Houston, Texas
- Argentina (4):
  - Buenos Aires, Capital Ferderal
  - Buenos Aires
  - Ciudad de Bs As
  - Córdoba
- Australia (6):
  - Camperdown
  - Parkville
  - Randwick
  - Westmead
  - Woodville South
  - Woolloongabba
- Vienna, Austria
- Canada (3):
  - London, Ontario
  - Cote Du Palais, Quebec
  - Montreal, Quebec
- Chile (4):
  - Puente Alto
  - Santiago
  - Talca
  - Viña del Mar
- Nicosia, Cyprus
- France (2):
  - Montpellier
  - Paris
- Münster, Germany
- Greece (2):
  - Athens
  - Thessaloniki
- Hungary (4):
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
- Italy (3):
  - Bari
  - Cagliari
  - Torino
- Oslo, Norway
- Portugal (3):
  - Carnaxide-lisboa
  - Coimbra
  - Lisbon
- Singapore, Singapore
- South Africa (2):
  - Cape Town
  - Johannesburg
- Spain (6):
  - Barcelona
  - La Coruã'a
  - La Laguna / Santa Cruz de Tenerife
  - Madrid
  - Santander
  - Valencia
- Uppsala, Sweden
- Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Antalya
  - Istanbul
  - Izmir
- United Kingdom (3):
  - Glasgow
  - Leicester
  - Manchester

REFERENCES:
- [Derived] Flechner SM, Gurkan A, Hartmann A, Legendre CM, Russ GR, Campistol JM, Schena FP, Hahn CM, Li H, Korth-Bradley JM, Tai SS, Schulman SL. A randomized, open-label study of sirolimus versus cyclosporine in primary de novo renal allograft recipients. Transplantation. 2013 May 27;95(10):1233-41. doi: 10.1097/TP.0b013e318291a269. PMID 23689085